CLINICAL TRIAL: NCT04283851
Title: Dynamic Parameters in Evaluation of Fluid Resposiveness in Cardiac Surgery Patients in the Early Postoperative Period
Brief Title: Dynamic Parameters in Evaluation of Fluid Responsiveness
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Martin Balik, Principal Investigator: Jan Horejsek, General University Hospital in Prague, Charles University, Czech Republic
Other Study IDs: 992/19 S-IV
Record Dates: First submitted 2020-01-27; First posted 2020-02-25 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Hypovolemia; Hypotension; Surgery
Keywords: fluid responsiveness; fluid administration; volume expansion; end-expiratory occlusion test; end-inspiratory occlusion test; diastolic parameters of cardiac ventricles; echocardiography; heart-lung interactions
MeSH Terms: conditions — Hypovolemia; Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: testing functional haemodynamic parameters for preload assessment — dynamic testing of preload responsivity plus echocardiography

SUMMARY:
Intravenous infusion of fluids in patients after surgery is a very important part of treatment. However, administering too much or too little fluid can lengthen the stay in the intensive care unit or even harm the patient. Therefore, fluid therapy should be tailored to the individual needs of each patient. Several methods are available to assess which patients will likely benefit from fluid administration. However, each of these methods is useful only under certain conditions. The study aims to explore some less-known, yet promising tests which could make adequate fluid administration more precise and easier to achieve.

DETAILED DESCRIPTION:
Adequate fluid therapy is one of the most important variables influencing patient outcome in intensive care. Fluid therapy should be tailored to the individual needs of each patient. Static parameters of preload have proved to be of little predictive value, therefore dynamic parameters are preferred for prediction of fluid responsiveness. Ideally, the cardiac output increases by 10% after a standardised fluid challenge. There are several methods already available to differentiate fluid-responsive from fluid-unresponsive patients, most notably the passive leg-raise. However, each of these methods has its own set of indications and contraindications. Also, a combination of tests could guide clinician´s decision in cases where the results of a single test are not entirely conclusive. Therefore, it would be desirable to add some less-known methods for prediction of fluid responsiveness, like the end-expiratory and end-inspiratory occlusion tests along with the assessment of diastolic properties of cardiac ventricles.

The aims of the study are:

* to determine the optimal increase in LVOT VTi to reliably predict fluid responsiveness
* to explore the accuracy of echocardiographic LVOT VTi evaluation during end-expiratory and end-inspiratory occlusion tests and their combination
* to assess the difference in echocardiographic properties of cardiac ventricles in fluid-responsive and fluid-unresponsive patients
* to compare the prediction based on echocardiography with the response to a standardised fluid challenge
* to assess the feasibility and practicality of echocardiographic monitoring in anesthetised cardiac surgery patients in intensive care

ELIGIBILITY:
Inclusion Criteria:

* patients after elective coronary artery bypass grafting
* hypovolemia indicated for volumotherapy by the attending physician based on clinical and laboratory signs (ScvO2 under 65 % with serum lactate above 2 mmol/l, increase of vasopressoric support with CVP under 5 mmHg)
* intubated and ventilated patients
* sedation without spontaneous breathing activity
* no pulmonary pathology on X-ray after surgery
* normal systolic and diastolic function of both ventricles (left ventricular ejection fraction above 50 %, TAPSE of the right ventricle above 20 mm, FAC of the right ventricle above 30 %)
* informed consent signed before surgery

Exclusion Criteria:

* aggresive artificial ventilation (PEEP above 10 cmH2O, Pmax above 30 cm H2O)
* ARDS, pneumothorax, fluidothorax
* hemodynamically significant valvular disease
* atrial fibrillation or other arrhythmia with irregular heartbeat
* intraabdominal hypertension with pressures above 15 mmHg
* open thorax
* bad echogenicity

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients undergoing elective CABG at the Deparment of Cardiovascular Surgery of the General University Hospital in Prague, who meet all the inclusion criteria and give their informed consent.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Prediction of fluid responsiveness | The first hour after surgery
  fluid responsiveness is defined as a 10 % increase in cardiac output after a standardised fluid challenge; the prediction will be made based on the diastolic properties of both cardiac ventricles and the changes in LVOT VTi during end-expiratory and end-inspiratory occlusion tests

SECONDARY OUTCOMES:
Echocardiographic evaluation of LVOT VTi and its changes | The first hour after surgery
  TTE measurement of LVOT VTi and its changes during end-expiratory, end-inspiratory occlusion tests and after a standardised fluid challenge of a colloid
Cardiac output monitoring with Vigileo FloTrac | The first hour after surgery
  continous measurement of cardiac output with Vigileo FloTrac and its correlation with the changes of echocardiographic parameters
Arterial pressure response | The first hour after surgery
  invasive arterial blood pressure
Heart rate response | The first hour after surgery
  heart rate
Oxygenation response | The first hour after surgery
  pulse oxymetry
Central venous pressure response | The first hour after surgery
  central venous pressure

CONTACTS AND LOCATIONS:
Overall Officials: Michal Porizka, MD, PhD, Study Director — Dept of Anest and Intensive Care, General University Hospital, Prague
Locations (1):
- Dept of Anaesthesia and Intensive Care, General University Hospital, 1st Medical Faculty, Charles University, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Georges D, de Courson H, Lanchon R, Sesay M, Nouette-Gaulain K, Biais M. End-expiratory occlusion maneuver to predict fluid responsiveness in the intensive care unit: an echocardiographic study. Crit Care. 2018 Feb 8;22(1):32. doi: 10.1186/s13054-017-1938-0. PMID 29415773
- [Background] Monnet X, Marik PE, Teboul JL. Prediction of fluid responsiveness: an update. Ann Intensive Care. 2016 Dec;6(1):111. doi: 10.1186/s13613-016-0216-7. Epub 2016 Nov 17. PMID 27858374
- [Background] Monnet X, Bleibtreu A, Ferre A, Dres M, Gharbi R, Richard C, Teboul JL. Passive leg-raising and end-expiratory occlusion tests perform better than pulse pressure variation in patients with low respiratory system compliance. Crit Care Med. 2012 Jan;40(1):152-7. doi: 10.1097/CCM.0b013e31822f08d7. PMID 21926581
- [Background] Monnet X, Osman D, Ridel C, Lamia B, Richard C, Teboul JL. Predicting volume responsiveness by using the end-expiratory occlusion in mechanically ventilated intensive care unit patients. Crit Care Med. 2009 Mar;37(3):951-6. doi: 10.1097/CCM.0b013e3181968fe1. PMID 19237902
- [Background] Marques NR, De Riese J, Yelverton BC, McQuitty C, Jupiter D, Willmann K, Salter M, Kinsky M, Johnston WE. Diastolic Function and Peripheral Venous Pressure as Indices for Fluid Responsiveness in Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2019 Aug;33(8):2208-2215. doi: 10.1053/j.jvca.2019.01.007. Epub 2019 Jan 4. PMID 30738752
- [Background] Pagourelias ED, Efthimiadis GK, Parcharidou DG, Gossios TD, Kamperidis V, Karoulas T, Karvounis H, Styliadis IH. Prognostic value of right ventricular diastolic function indices in hypertrophic cardiomyopathy. Eur J Echocardiogr. 2011 Nov;12(11):809-17. doi: 10.1093/ejechocard/jer126. Epub 2011 Aug 15. PMID 21846651
- [Result] Jozwiak M, Depret F, Teboul JL, Alphonsine JE, Lai C, Richard C, Monnet X. Predicting Fluid Responsiveness in Critically Ill Patients by Using Combined End-Expiratory and End-Inspiratory Occlusions With Echocardiography. Crit Care Med. 2017 Nov;45(11):e1131-e1138. doi: 10.1097/CCM.0000000000002704. PMID 28857907